CLINICAL TRIAL: NCT05711940
Title: A Phase III, Multicentre, Randomised, Double-blind, Controlled Study to Investigate the Efficacy, Safety, and Tolerability of Two Administrations of COMP360 in Participants With Treatment-resistant Depression
Brief Title: Efficacy, Safety, and Tolerability of Two Administrations of COMP360 in Participants With TRD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMP 006
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: psilocybin
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 25 mg COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- 10 mg COMP360 Psilocybin (Experimental): 10 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- 1 mg COMP360 Psilocybin (Active Comparator): 1 mg COMP360 Psilocybin, active comparator
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — COMP360 Psilocybin administered under supportive conditions
  Other Names: COMP360

SUMMARY:
Efficacy, Safety, and Tolerability of two administrations of COMP360 in participants with treatment-resistant depression (TRD)

DETAILED DESCRIPTION:
This is a phase III, international, multi-centre, randomised, parallel group, fixed repeat dose, double-blind, controlled study. The study population will include participants aged ≥18 years with TRD.

Overall, 568 participants are to be randomised in a 2:1:1 ratio to receive COMP360 25 mg, 10 mg or 1 mg.

The study comprises three parts (A, B, and C) and will last approximately 62 weeks including a three- to ten-week screening period.

Part A will include a nine-week follow-up from initial investigational product (IP) administration.

Part B will include a further 17 weeks follow-up out to 26 weeks from initial IP administration.

Part C will include a further 26 weeks follow-up out to 52 weeks from initial IP administration.

In this study, the aim is to assess the efficacy of COMP360, administered with psychological support in adult participants with TRD, in improving symptoms of depression.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged ≥18 years at Screening
2. Major depression without psychotic features (single or recurrent episode as informed by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-5])
3. If the current major depressive episode is the participant's first lifetime episode of depression, the length of the current episode must be ≥3 months and ≤2 years at Screening
4. MADRS total score ≥20 at Screening and Baseline to ensure at least moderate severity of depression
5. TRD, defined as failure to respond to an adequate dose and duration of two, three, or four different pharmacological treatments for the current episode as determined through the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and using the supplementary advice on additional antidepressants not included in MGH-ATRQ
6. At Screening, agreement to discontinue all prohibited medications

Key Exclusion Criteria:

1. Prior or ongoing bipolar disorder, any psychotic disorder, including schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder (unless substance induced or due to a medical condition), antisocial personality disorder as assessed by a structured clinical interview (MINI 7.0.2)
2. Lifetime paranoid, schizoid, schizotypal, histrionic, narcissistic personality disorder, or any ongoing serious psychiatric comorbidity based on medical history and clinical judgement
3. Borderline personality disorder as demonstrated by medical history or the Mini International Neuropsychiatric Interview Plus (MINI plus) - borderline personality disorder module
4. Ongoing post-traumatic stress disorder, obsessive-compulsive disorder, or anorexia nervosa as assessed by medical history and a structured clinical interview (MINI 7.0.2)
5. Psychiatric inpatient within the past 12 months prior to Screening
6. Use of electroconvulsive therapy, deep brain stimulation, or vagus nerve stimulation during the current depressive episode
7. Transcranial magnetic stimulation within the past six months prior to Screening
8. Current enrolment in a psychological therapy programme that will not remain stable for the duration of the study. Psychological therapies cannot have been initiated within 30 days prior to Screening
9. Exposure to COMP360 psilocybin therapy prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
COMP360 25 mg versus COMP360 1 mg for the change from baseline in MADRS total score. | Week 6
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity

SECONDARY OUTCOMES:
COMP360 25 mg versus COMP360 1 mg for the change from baseline in Sheehan Disability Scale (SDS) total score. | Week 6
  Sheehan Disability Scale (SDS) is a brief, five-item self report inventory that assesses functional impairment in work/school, social life, and family life.
COMP360 25 mg versus COMP360 10 mg for the change from baseline in MADRS total score. | Week 6
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity
COMP360 25 mg versus COMP360 10 mg for the change from baseline in Sheehan Disability Scale (SDS) total score. | Week 6
  Sheehan Disability Scale (SDS) is a brief, five-item self report inventory that assesses functional impairment in work/school, social life, and family life.

CONTACTS AND LOCATIONS:
Locations (116):
- United States (62):
  - Lighthouse Psychiatry Scottsdale, Gilbert, Arizona
  - Clinical Innovations, Inc., Bellflower, California
  - M3 Wake Research, Encino, California
  - The Regents of the University of California - San Diego, La Jolla, California
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - CalNeuro Research Group, Inc, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Piedmont Hospital Neuroscience Centre, Oakland, California
  - ATP Clinical Research, Inc., Orange, California
  - CITrials, Riverside, California
  - Lumos Clinical Research Center, San Jose, California
  - Syrentis Clinical Research, Santa Ana, California
  - Stanford University, Stanford, California
  - ASCLEPES Research Centers, Thousand Oaks, California
  - Pacific Clinical Research Management Group, LLC, Upland, California
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Central Miami Medical Institute, LLC, Miami, Florida
  - Behavioral Clinical Research, Inc., Miami Lakes, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Clinical Neurosciecne Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - APG Research, LLC- Advanced Psychiatric Group, Orlando, Florida
  - University South Florida, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Psychiatric Medicine Associates, Skokie, Illinois
  - Harvard Medical School - McLean Hospital, Belmont, Massachusetts
  - Adams Clinical - Boston (Copley Clinical), Boston, Massachusetts
  - University of Massachusetts Medical School, North Worcester, Massachusetts
  - Adams Clinical - Boston, Watertown, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - University Of Michigan Comprehensive Depression Center, Ann Arbor, Michigan
  - Institute for Integrative Therapies, Eden Prairie, Minnesota
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC., Lincoln, Nebraska
  - Hassman Research Institute, Berlin, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - Fieve Clinical Research, Inc, New York, New York
  - Spectrum Neuroscience and Treatment Institute, New York, New York
  - Adams Clinical - New York, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Adams Clinical - New York, The Bronx, New York
  - University of Cincinnati, Department of Psychiatry & Behavirol Neuroscience, Cincinnati, Ohio
  - Cleveland Clinic - Lutheran Hospital, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - The University of Texas at Austin - Dell Medical School, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - Center for Depression Research and Clinical Care, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Brain Health Consultants and TMS Center, Houston, Texas
  - HCA Healthcare Research Institute - Medical City Green Oaks Hospital, Plano, Texas
  - Cedar Clinical Research, Draper, Utah
  - The University of Utah - Huntsman Mental Health Institute, Salt Lake City, Utah
  - Seattle Neuropsychiatric Treatment Center, Seattle, Washington
- Canada (9):
  - Diex Recherche Sherbrooke Inc., Québec, B.C.
  - Medical Arts Health Research Centre, Kamloops, Kamloops, British Columbia
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Medical Arts Research Group - Penticton, Penticton, British Columbia
  - Chatham-Kent Clnical Trials Centre, Chatham, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Centre for Neurology Studies, Vancouver
  - Medical Arts Research Group, Vancouver
- Czechia (6):
  - National Institute of Mental Health, Klecany
  - Neuroterapie KH Sro, Kutná Hora
  - Psychiatric Ambulance, Ostrava
  - A-Shine s.r.o., Pilsen
  - Psychedelicka klinika, s.r.o., Prague
  - Institut Neuropsychiatricke Pece, Prague
- Aalborg Universitetshospital-Psykiatrien Region Nordjylland, Aalborg, Denmark
- France (4):
  - Centre Hospitalier Universitaire de Nimes (CHU) - Hopital Universitaire Caremeau, Nîmes
  - Universite Paris VI Pierre et Marie Curie - Hopital de La Salpetriere - Centre Emotion - USR 3246 (CNRS UMR 7593), Paris
  - Centre Hospitalier Sainte Anne - Clinique des Maladies Mentales et de l'Encephale (CMME), Paris
  - Ghu-Centre Hospitalier Sainte Anne, Centre de Recherche Clinique, Paris
- Germany (3):
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Johann Wolfgang Goethe-Universitaet Frankfurt am Main - Klinik fuer Psychiatrie, Psychosomatik und Psychotherapie, Frankfurt
  - ZiP Campus Luebeck, Lübeck
- Ireland (2):
  - Tallaght University Hospital, Dublin
  - La Nua Day Hospital Mental Health Centre, Galway
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leids Universitair Medisch Centrum (LUMC) (Leiden University Medical Center) - Leiden Institute for Brain and Cognition (LIBC), Leiden
  - Universitair Medisch Centrum Utrecht (UMC Utrecht), Utrecht
- Poland (3):
  - Promente - Ośrodek Badań Klinicznych, Bydgoszcz
  - Uniwersyteckle Centrum Kliniczne, Klinika Psychiatrii Doroslych, Gdansk
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Parc Sanitari Sant Joan de Deu (Sant Joan de Deu Serveis de Salut Mental), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - FIDMAG Hermanas Hospitalarias, Sant Boi de Llobregat
  - Hospital Universitario Río Hortega de Valladolid, Valladolid
  - Hospital Provincial de Zamora - Servicio de Psiquiatria, Zamora
- Sweden (4):
  - Vuxenpsykiatrimottagningen, Landskrona
  - Lunds Universitet - Medicinska Fakulteten (Lund University Faculty of Medicine), Lund
  - ClinSmart Sweden AB, Solna
  - Hälsoklustret, Stockholm
- United Kingdom (13):
  - Cornwall Partnership NHS Foundation Trust, Bodmin, Cornwall
  - Abraham Cowley Unit - Surrey and Borders Partnership NHS Foundation Trust, Chertsey
  - St. Pancras Clinical Research, Chester
  - Grounded Research Hub - Rotherham Doncaster & South Humber NHS Foundation Trust, Doncaster
  - Clinical Research Facility, Royal Devon and Exeter Hospital, Exeter
  - Fulbourn Hospital - Cambridgeshire And Peterborough NHS Foundation Trust, Fulbourn
  - St. Pancras Clinical Research, London
  - King's College London - Institute of Psychiatry, Psychology, London
  - Clerkenwell Health, London
  - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust - Wolfson Research Centre, Newcastle
  - University Of Nottingham/Nottinghamshire Healthcare Trust, Institute Of Mental Health, Nottingham
  - The Warneford Hospital- NIHR Clinical Research Facility, Oxford
  - Sheffield Health and Social Care NHS Foundation Trust, Sheffield